CLINICAL TRIAL: NCT00415857
Title: Potential of Immunotherapy to Convert a Complete Cytogenetic Remission in Chronic Myelogenous Leukemia to a Molecular Complete Remission: Randomized Phase II Study of Proteinase 3 PR1 Peptide Mixed With Montanide ISA-51 VG Adjuvant and Administered With GM-CSF and Peginterferon Alfa-2b [PEG-INTRON(R), Schering Corporation]
Brief Title: Proteinase 3 PR1 Peptide Mixed With Montanide ISA-51 VG Adjuvant and Administered With GM-CSF and PEG-INTRON(R)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Vaccine sponsor ceased operations.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: The Vaccine Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0360
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Leukemia
Keywords: Chronic Myelogenous Leukemia; Leukemia; Peptide Vaccine; PR1 Peptide; Imatinib; Gleevec; GM-CSF; Sargramostim; Leukine; Peginterferon alfa-2b; Peg-Intron
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Protein Subunit Vaccines; peginterferon alfa-2b; Imatinib Mesylate; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PR1 + Imatinib (Experimental): PR1 peptide will be administered at a dose of 0.5 mg of PR1 on weeks 0, 3, 6 and 18 for a total of 4 doses. Continue receiving imatinib by mouth at the same dose received during the last 6 months. GM-CSF 75 micrograms subcutaneously in the same area as the vaccine with every vaccination.
  Interventions: Biological: Peptide Vaccine (PR1 Peptide); Drug: Imatinib; Drug: GM-CSF
- PR1 + Imatinib + Interferon (Experimental): PR1 peptide will be administered at a dose of 0.5 mg of PR1 on weeks 0, 3, 6 and 18 for a total of 4 doses. Subcutaneous injection of interferon 0.5 microg/kg with each PR1 vaccination. GM-CSF 75 micrograms subcutaneously in the same area as the vaccine with every vaccination.
  Interventions: Biological: Peptide Vaccine (PR1 Peptide); Drug: Peginterferon alfa-2b; Drug: Imatinib; Drug: GM-CSF

INTERVENTIONS:
Biological: Peptide Vaccine (PR1 Peptide) — PR1 peptide will be administered at a dose of 0.5 mg of PR1 on weeks 0, 3, 6 and 18 for a total of 4 doses.
  Other Names: PR1 Vaccine
Drug: Peginterferon alfa-2b — Subcutaneous injection of interferon 0.5 microg/kg with each PR1 vaccination.
  Other Names: Peg-Intron
  Arms: PR1 + Imatinib + Interferon
Drug: Imatinib — Continue receiving imatinib by mouth at the same dose received during the last 6 months.
  Other Names: Gleevec
Drug: GM-CSF — 75 micrograms subcutaneously in the same area as the vaccine with every vaccination.
  Other Names: Sargramostim; LeukineTM

SUMMARY:
The goal of this clinical research study is to find out if using the PR1 peptide vaccine (PR1) without PEG-Intron® (interferon) or in combination with interferon can reduce or eliminate disease in patients who have CML that is in cytogenetic remission after treatment with imatinib mesylate, but who still have small amounts of disease able to be noticed (detected). Researchers want to see if giving low doses of interferon together with PR1 may make the vaccine more effective. The safety of treatment in this study will also be studied.

DETAILED DESCRIPTION:
Your disease responded well to treatment with imatinib mesylate. It is in complete cytogenetic remission. This means that the Philadelphia chromosome (Ph), a change in genetic material that is believed to lead to leukemia, is no longer detectable (by the standard chromosome analysis) in your bone marrow and blood cells. A molecular remission, which is what researchers want you to achieve, means a greater reduction or a complete elimination of the Ph.

The small amounts of disease can be detected using a technique called polymerase chain reaction (PCR). This is a very powerful test that can detect very small amounts of disease that can still be present in the bone marrow and/or blood cells.

PR1 is an experimental vaccine made from a protein that is found in large amounts in leukemia cells in CML.

Imatinib mesylate (which you are already receiving as standard therapy) is designed to bind to certain proteins on the tumor cells, which may prevent the cells from growing.

Interferon is a drug that was used as standard therapy for patients with CML before imatinib mesylate was available. It can help the immune system to function more effectively (causing leukemia cells to show more PR1), which may make leukemia cells a better target to be killed.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate). You will have your complete medical history recorded. You will have blood drawn (about 2 tablespoons) for routine tests. Women who are able to have children must have a negative blood (about 1 teaspoon) or urine pregnancy test. You will also have blood drawn (about 1 tablespoon) to see if you have the necessary protein (called HLA-A2) needed for the vaccine to recognize your cells. You will also have additional blood drawn (about 1 tablespoon) to test (using the PCR test) the levels of leukemia in your blood. You will have a bone marrow aspiration. To collect a bone marrow aspiration, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. You will have a chromosome test done on the number of chromosomes in your bone marrow (collected from your bone marrow aspiration). You will not have an additional procedure performed on you for this test. For this test, all of your chromosomes in 20 cells in your bone marrow will be counted to see if there may be any unhealthy changes (such as the Ph) present as well as how many may be present.

If you are found to be eligible to take part in this study, you will receive PR1 through a small needle just under your skin (subcutaneous injection). Imatinib mesylate will continue to be given to you by mouth at the dose that you are taking now as part of your standard therapy. PR1 will be mixed with a substance called Montanide ISA 51 VG, which is a regular procedure that will help your immune system respond to PR1.

You will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. Participants in one group will receive a subcutaneous injection of interferon with each PR1 vaccination. Participants in the other group will receive PR1 vaccination without interferon.

Regardless of what group you are assigned to, you will also receive, with each PR1 vaccination, a growth hormone called GM-CSF. The purpose of GM-CSF is to boost your immune system (in response to the PR1 vaccine) to help kill your leukemia. It is given as a subcutaneous injection in your arms or your thighs.

All participants will receive a total of 4 doses of the PR1 vaccine. The first 3 vaccinations are given every 3 weeks, and the last vaccination is given 18 weeks after the start of therapy in this study. You will receive all of these vaccinations at M. D. Anderson.

Every time you come in for an injection of PR1, you will have a physical exam, including measurement of your vital signs. You will have blood drawn (about 2 tablespoons) for routine tests, and you will have blood drawn (about 1 tablespoon) for the PCR test. After you receive the last vaccination, you will continue having the PCR test every 3 months to test the level of leukemia in your blood and to see if your disease is responding to the vaccine. You will have a bone marrow aspiration at 1 month and 6 months after the last vaccination. To measure the response of your immune system to PR1, blood will be drawn (about 2 tablespoons each) before the first vaccination, at Weeks 6, 18, 22 and 6 months after treatment.

You will be taken off this study if intolerable side effects occur or your disease progresses (comes out of remission).

This is an investigational study. PR1 mixed with Montanide ISA-51 VG is authorized by the FDA for use in research only. Interferon and GM-CSF are FDA-approved and commercially available. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/= 18 years with Philadelphia chromosome (Ph)- or BCR/ABLpositive CML (as determined by cytogenetics, FISH, or PCR).
2. Patients must have received imatinib therapy for at least 18 months and not have increased their dose of imatinib in the last 6 months.
3. Patients must be in complete cytogenetic remission.
4. Patients must have detectable BCR-ABL transcript levels meeting at least one of the following criteria: 1) Patient has never achieved a major molecular response (i.e., never reached levels <0.05%), and transcript levels have shown in at least two consecutive measures separated by at least 1 month to have increased by any value, or
5. continued from above: 2) Achieved a major molecular response that has been lost with an increase in transcript levels by at least 1-log over two consecutive analyses separated by at least 1 month, or 3) BCR-ABL transcript levels have reached a plateau defined as a ratio that is not more than 0.25-log (one fourth of a log) lower than the lowest value obtained in the last at least 6 months, with at least 2 values obtained during this period.
6. Patients must not have had a continuous interruption of imatinib therapy of greater than 14 days or any interruptions totaling 6 weeks within the 6 months prior to enrollment.
7. Patients must be HLA-A2 positive at one allele
8. Patients must give informed consent and sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.
9. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
10. Adequate organ function defined as: bilirubin <2 times upper limit of normal (ULN), creatinine <1.5 times ULN, and serum glutamate pyruvate transaminase (sGPT) <2.5 times ULN.
11. Women of childbearing potential should practice effective methods of contraception.

Exclusion Criteria:

1. Patients with a history or clinical evidence of autoimmune disorders
2. Patients receiving immunosuppressive therapy including cyclosporine, or FK506 within 3 months of study entry
3. Chronic use (> 2 weeks) of greater than physiologic doses of corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 28 days of the first day of study drug treatment (topical and inhaled corticosteroids are permitted)
4. GM-CSF or interferon administration within 1 month of first PR1 injection
5. Patients receiving any other investigational agents currently or within the past 4 weeks. Patients must have recovered from any adverse effects of investigational therapy.
6. Patients who are pregnant or breast-feeding
7. Patients with clinically significant heart disease (New York Heart Association (NYHA) Class III or IV)
8. Patients with positive cANCA
9. History of HIV positivity or AIDS
10. Chloroma at time of study screening
11. Prior vaccine therapy for Chronic myelogenous leukemia (CML)
12. Known allergy to Montanide ISA-51 VG adjuvant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: December 20, 2006 to March 13, 2009. All recruitment done at the University of Texas (UT) MD Anderson Center.
Pre-assignment Details: Due to the unavailability of the study drug (vaccine) enrollment was halted and the study eventually terminated when additional attempts were unsuccessful to obtain a supply of vaccine.
Groups:
- PR1 + Imatinib: PR1 peptide administered dose 0.5 mg on weeks 0, 3, 6 and 18 for a total of 4 doses, with oral Imatinib at same dose received during last 6 months. Granulocyte-macrophage colony-stimulating factor (GM-CSF) 75 micrograms subcutaneously in same vaccine area with every vaccination.
- PR1 + Imatinib + Interferon: PR1 peptide administered dose 0.5 mg on weeks 0, 3, 6 and 18 for a total of 4 doses, with oral Imatinib at same dose received during last 6 months. Granulocyte-macrophage colony-stimulating factor (GM-CSF) 75 micrograms subcutaneously in same vaccine area with every vaccination, and Peginterferon alfa-2b 0.5 microg/kg subcutaneous injection with each PR1 vaccination.
Period: Overall Study
Arm/Group | PR1 + Imatinib | PR1 + Imatinib + Interferon
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PR1 + Imatinib | PR1 + Imatinib + Interferon | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: Years] | 45 [35 to 55] | 46 [29 to 50] | 46 [29 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Molecular Response Rate
Description: Molecular response rate is number of respondents compared to total participants. Molecular Response is defined as a greater than a one-log reduction of Breakpoint Cluster Region-Abelson Murine Leukemia (BCR-ABL) transcript levels by quantitative polymerase chain reaction (PCR) from the baseline level at the time vaccination was initiated, or a disappearance of BCR-ABL transcripts, as measured by reverse transcription polymerase chain reaction (RT-PCR), occurring within 6 months from the last vaccination. Participants receive a series of 4 vaccinations administered at 3-week intervals and the fourth (final) vaccination administered 3 months after the third vaccination with blood draw to test PCR following every 3 months to test the level of leukemia in the blood and to see if disease is responding to the vaccine.
Time Frame: Baseline to 18 weeks, up to 6 months post final vaccination for overall study participation period.
Measure: Number; unit: percentage of participants
Arm/Group | PR1 + Imatinib | PR1 + Imatinib + Interferon
Number analyzed (Participants) | 2 | 3
percentage of participants | 0 | 0

2. Secondary Outcome: Number of Participants With Immunologic Response
Description: Immunologic Response (immune response) is defined as an increase of ≥ 0.5 PR1-HLA-A2 [human leukocyte antigen-A2 (HLA-A2)] tetramer cells / μl at the time of either the 3rd or 4th vaccination compared to the pre study absolute PR1-HLA-A2 tetramer cells / μl. Participants receive a total of 4 vaccinations over a period of 18 weeks (i.e., one vaccination each on weeks 0, 3, 6, and 18). Participants assessed after 3rd and 4th vaccination for immunologic response.
Time Frame: Period of 18 weeks (i.e., one vaccination each on weeks 0, 3, 6, and 18).
Measure: Number; unit: participants
Arm/Group | PR1 + Imatinib | PR1 + Imatinib + Interferon
Number analyzed (Participants) | 2 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants followed for one month after removal from study. The overall study period was 1 years and 8 months.
Arm/Group | PR1 + Imatinib | PR1 + Imatinib + Interferon
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR1 + Imatinib (N=2) | PR1 + Imatinib + Interferon (N=3)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes